CLINICAL TRIAL: NCT00087282
Title: A Non-Randomized Phase II Study of Sequential Irinotecan (CPT-11) And Flavopiridol In Patients With Advanced Hepatoma
Brief Title: Irinotecan and Flavopiridol in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000373877; MSKCC-04038; NCI-6475
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — alvocidib; Irinotecan

INTERVENTIONS:
Drug: alvocidib
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and flavopiridol, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with flavopiridol works in treating patients with advanced liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with advanced hepatocellular carcinoma treated with irinotecan and flavopiridol.

Secondary

* Determine the response rate and overall survival in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is an open-label, non-randomized study.

Patients receive irinotecan IV over 30 minutes and flavopiridol IV over 1 hour on days 1, 8, 15, and 22. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 16-32 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma

  * Advanced disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Prior local therapy (e.g., surgery, hepatic arterial embolization, radiofrequency ablation, or cryoablation) allowed provided therapy was completed ≥ 8 weeks before study entry AND ≥ 1 of the following conditions are met:

  * Target lesion was not subjected to local therapy
  * 25% increase in the size of target lesion within the field of prior local therapy

    * Lesions treated with external beam radiotherapy are not acceptable as target lesions
* Child-Pugh class A or B status if liver cirrhosis is present

  * Score 7 or 8 only
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* See Disease Characteristics
* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No deep vein thrombosis within the past 6 months

  * Patients maintained on anticoagulation therapy for an event that occurred more than 6 months ago are eligible
* No myocardial infarction within the past 6 months
* No cardiac arrhythmia within the past 6 months

  * Rate-controlled atrial fibrillation allowed if stable for at least 6 months

Pulmonary

* No pulmonary embolus within the past 6 months

  * Patients maintained on anticoagulation therapy for an event that occurred more than 6 months ago are eligible

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to flavopiridol or irinotecan
* No clinically significant gastrointestinal bleeding requiring hospitalization within the past month
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other malignancy within the past 3 years except carcinoma in situ of the cervix, adequately treated basal cell skin cancer, or superficial bladder tumors [Ta, Tis, or T1]

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior systemic biologic therapy

Chemotherapy

* No prior systemic chemotherapy for hepatocellular carcinoma
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* No prior organ allograft

Other

* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent vitamins, antioxidants, or herbal preparations and supplements

  * Single-tablet multivitamin allowed
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Abou-Alfa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Gary K. Schwartz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States